CLINICAL TRIAL: NCT05054920
Title: Eccentric Versus Concentric Exercises for Rotator Cuff Tendinopathy in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Badr University (Other)
Responsible Party: Principal Investigator, Mina Magdy Wahba, Assistant lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mina
Record Dates: First submitted 2021-09-19; First posted 2021-09-23 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis; Rotator Cuff Tendinosis; Tendinopathy
MeSH Terms: conditions — Arthritis, Rheumatoid; Rotator Cuff Injuries; Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentric exercises group (Experimental): patient will do Concentric exercises. Patients will receive 3 sessions per week for 4 weeks. Exercise will be done under the supervision of the same physical therapist. During each session.
  Exercise will be in the form of glenohumeral scaption, internal and external rotation exercises.
  patient will also do stretching for posterior capsule and pectoralis minor
  Interventions: Other: concentric exercises; Other: Stretching
- Eccentric exercises group (Experimental): patient will do eccentric exercises. Patients will receive 3 sessions per week for 4 weeks. Exercise will be done under the supervision of the same physical therapist during each session.
  Exercise will be in the form of glenohumeral scaption, internal and external rotation exercises.
  patient will also do stretching for posterior capsule and pectoralis minor
  Interventions: Other: eccentric exercises; Other: Stretching

INTERVENTIONS:
Other: concentric exercises — concentric exercises for rotator cuff. internal rotators, external rotators and abductors Patient will do 3 sets of 10 repetitions resistance will be personalized to each patients
  Arms: Concentric exercises group
Other: eccentric exercises — Eccentric exercises exercises for rotator cuff internal rotators, external rotators and abductors Patient will do 3 sets of 10 repetitions resistance will be personalized to each patients
  Arms: Eccentric exercises group
Other: Stretching — stretching exercise for posterior capsule and pectoralis minor each stretch will be done for 30 seconds and repeated 3 times

SUMMARY:
Study aiming at determining the efficacy of eccentric versus concentric exercises for improving tendon biological characteristics, pain, and shoulder overall function for rotator cuff tendinopathy in patients with Rheumatoid arthritis (RA).

Moreover, investigation the relationship between RA activity and the severity of rotator cuff tendinopathy.

Patients will be randomly assigned into either concentric or eccentric exercise group. Randomizations will be done using computer random generated numbers.

DETAILED DESCRIPTION:
Study aiming at determining the efficacy of eccentric versus concentric exercises for improving tendon biological characteristics, pain, and shoulder overall function for rotator cuff tendinopathy in patients with RA. Moreover, investigation the relationship between RA activity and the severity of rotator cuff tendinopathy.

Patients will be randomizations using computer random generated numbers. patients will receive either eccentric or concentric exercises for internal, external rotators and abductors muscles All patient will do stretching for posterior capsule and pectoralis minor Tendon biological changes and subacromial space will be assessed using musculoskeletal ultrasonography Shoulder function will be assessed using SPADI (shoulder pain and disability index Pain will be assessed using Visual Analogue Scale (VAS) Rheumatoid arthritis disease activity will be assessed using Disease Activity Score-28 for Rheumatoid Arthritis with erythrocyte sedimentation rate (DAS 28 ESR) patient will be assessed at base-line and after finishing of the study

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients diagnosed with RA according to 2010 (American College of Rheumatology)(ACR)/European League Against Rheumatism (EULAR) Classification Criteria for RA
2. Patients diagnosed with rotator cuff tendinopathy based on clinical and musculoskeletal Ultrasonography (MSUS) finding.
3. Patient complaining of shoulder pain for at least 3 months
4. Positive jobs test or hornblower sign or left off test
5. Age ranged from 18 to 50 years.

Exclusion Criteria:

1. Patient indicated for surgical repair of rotator cuff
2. Patient with previous shoulder surgery.
3. Patient with history of intra-articular shoulder fracture.
4. Patient with history of shoulder dislocation
5. Diabetes mellitus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Shoulder function | one month
  shoulder Pain and Disability Index (SPADI): It is a self-reported questionnaire evaluating the function of the shoulder.

SECONDARY OUTCOMES:
tendon thickness, fibrillar pattern and echogenicity | one month
  tendon thickness, fibrillar pattern and echogenicity as measured Ultrasonography
subacromial space | one month
  shoulder subacromial space as measured by Ultrasonography
Pain measured by Visual analogue scale (VAS) | one month
  pain as measured by Visual analogue scale which a 10 cm scale marked at the beginning zero indicating no pain and 10 at the end indicating worst pain
ESR | one month
  Erythrocyte sedimentation rate
disease activity score 28 Erythrocyte sedimentation rate (DAS 28- ESR) | one month
  disease activity score 28 Erythrocyte sedimentation rate High disease activity is defined as a DAS 28 ESR>5.1, moderate activity as a DAS 28 ESR between 3.2 and ≤5.1, low activity as a DAS 28 ESR between 3.2 and >2.6, and remission as a DAS 28 ESR less than 2.6

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Shawki Abdelsalam, PhD, Study Chair — Assistance Professor,Faculty of Physical Therapy Cairo University; Mona Fagaal, PhD, Study Director — Assistance Professor, Faculty of Physical Therapy Badr University in Cairo; Mohammed Moustafa Aldosouki Hegazy, PhD, Study Director — Lecturer,Faculty of Physical Therapy Cairo University; Rasmia Mohamed Hassan ElGohry, phD, Study Director — Cairo University
Locations (1):
- Badr University in Cairo (BUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No